CLINICAL TRIAL: NCT03047655
Title: Effects of Short-term Interventions for a Healthy Lifestyle on the Human Lipidome in Subjects With Metabolic Syndrome
Acronym: GesundLeben
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Institute of Human Nutrition (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Director (Dpt. Clinical Nutrition), German Institute of Human Nutrition
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GesundLeben
Record Dates: First submitted 2016-11-21; First posted 2017-02-09 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Metabolic Syndrome; NAFLD; Obesity; Hypertension
MeSH Terms: conditions — Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Obesity; Hypertension | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity only (Active Comparator): pedometers have to be used throughout all days; daily amount of steps is reported via App or website; 10000 steps are defined as daily goal
  Interventions: Behavioral: Lifestyle intervention (physical activity)
- Physical activity + Dietary treatment (Active Comparator): pedometers have to be used throughout all days; daily amount of steps is reported via App or website; 10000 steps are defined as daily goal
  additionally, subjects will be provided with one healthy muffin per day (450 kcal; low GI, high load of PUFA and isomaltulose) over 6 weeks
  Interventions: Behavioral: Lifestyle intervention (physical activity); Dietary Supplement: Lifestyle intervention (PUFA/isomaltulose-enriched muffin)

INTERVENTIONS:
Behavioral: Lifestyle intervention (physical activity) — Dietary treatment with or without additional motivation on more physical activity
Dietary Supplement: Lifestyle intervention (PUFA/isomaltulose-enriched muffin)
  Arms: Physical activity + Dietary treatment

SUMMARY:
A growing number of cross-sectional studies is investigated the role of the human lipidome as a new biomarker for metabolic diseases. However, data on this issue is still sparse and especially interventional data is not available up to now.

"GesundLeben" will provide data on 100 human subjects with metabolic syndrome, undergoing distinct types of lifestyle intervention for 6 weeks. Standardized metabolic assessment will be covered with routine laboratory parameters and oral glucose tolerance test as well as non-radiologic anthropometric measurements.

DETAILED DESCRIPTION:
A growing number of cross-sectional studies is investigated the role of the human lipidome as a new biomarker for metabolic diseases. However, data on this issue is still sparse and especially interventional data is not available up to now. We intend to clarify, if the human lipidome is correlating with metabolic state and if changes in this state reflect on the lipidome. Using high-throughput shot-gun technique, we will be able to measure several hundreds of lipid species in one blood sample.

The "GesundLeben" trial will provide data on 100 human subjects with metabolic syndrome, undergoing distinct types of lifestyle intervention for 6 weeks. The cohort will be designed to include participants from both sexes, but be restricted on subjects without impaired glucose tolerance.

Standardized metabolic assessment will be covered with routine laboratory parameters (e.g. transaminases, HbA1c) and oral glucose tolerance test as well as non-radiologic anthropometric measurements (BMI, WHR, BIA).

ELIGIBILITY:
Inclusion Criteria:

* hypertension
* NAFLD
* obesity
* hyperuricemia
* dyslipoproteinemia

Exclusion Criteria:

* prediabetes / overt diabetes mellitus
* present cancer
* systemic infection
* chronic inflammatory disease
* recent stroke / myocardial infarction (6 months)
* pregnancy
* addiction / severe psychiatric diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-09 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
change in lipidome pattern | 6 weeks
  complex human lipidome (blood levels of several hundreds of lipid species) will be assessed before and after intervention
reduction of blood pressure | 6 weeks
  systolic and diastolic blood pressure
NAFLD reduction | 6 weeks
  NAFLD, estimated by fatty liver index (FLI)
weight loss | 6 weeks
  loss in body weight / BMI

SECONDARY OUTCOMES:
reduction of insulin resistance | 6 weeks
  assessed by oral glucose tolerance test, glucose and insulin levels; IS indices (Matsuda, IGI etc.)
improvement in quality of life | 6 weeks
  standardized questionnaires

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - German Institut for Human Nutrition; Department for Clinical Nutrition, Bergholz-Rehbrücke, Brandenburg
  - DIfE (German Institute for Human Nutrition), Berlin

IPD SHARING:
Plan to Share IPD: Undecided